CLINICAL TRIAL: NCT02771249
Title: Impact of Once-Weekly Rifapentine and Isoniazid on the Steady State Pharmacokinetics of Dolutegravir and Darunavir Boosted With Cobicistat in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160112; 16-CC-0112
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2021-12-28

CONDITIONS: HIV Infected Population With Latent Tuberculosis
Keywords: Fixed Sequence; Intrasubject Drug-Drug Interaction; Open-Label
MeSH Terms: interventions — cobicistat mixture with darunavir; Isoniazid; Pyridoxine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm B (Experimental): Arm B will be comprised of two phases: (1) DRV/c once daily alone (days 1-4) and (2) DRV/c once daily + RPT and INH once weekly (days 5-19).
  Interventions: Drug: rifapentene (RPT); Drug: darunavir/cobicistat (DRV/c); Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine

INTERVENTIONS:
Drug: rifapentene (RPT) — RPT is a long-acting rifamycin used in combination with INH in the treatment of LTBI.
Drug: darunavir/cobicistat (DRV/c) — DRV is a protease inhibitor (PI) indicated in the treatment of HIV infection.33 DRV requires coadministration with RTV (100 mg once or twice daily) or COBI (150 mg daily), the latter of which has been coformulated into a fixed-dose tablet with DRV (DRV/c 800/150 mg).
Drug: Isoniazid (INH) — INH is an antimycobacterial agent that can be used alone or in combination with RPT for the treatment of LTBI. Given with Pyridoxine (vitamin B6)
Dietary Supplement: Pyridoxine

SUMMARY:
People with human immunodeficiency virus (HIV) often take several medicines to control HIV. Dolutegravir and darunavir boosted with cobicistat are HIV medicines that people may take. They may also need to take medicines for an infection called latent tuberculosis (TB). Researchers think a once-weekly treatment for latent TB would be easier for people with HIV to take. This once weekly treatment consists of two drugs: rifapentine and isoniazid. However, they need to see how TB drugs and HIV drugs interact.

Objective:

To learn how anti-HIV and anti-TB drugs affect each other so that people taking these drugs together can be treated safely.

Eligibility:

Healthy adults ages 18 65.

Design:

Participants will be screened with a medical history and physical exam. They will have vital signs taken and give a blood sample. Women will have a pregnancy test.

Participants cannot take any other medicines during the study, including vitamins. Only occasional, infrequent use of acetaminophen (Tylenol , max 2000 mg/day), ibuprofen (Motrin or Advil ), naproxen (Aleve ), loperamide (Imodium ), and/or antihistamines (such as Benadryl , Zyrtec , Claritin , etc.) will be allowed.

Participants will be assigned to one of three groups. Each group will take a different study drug, once or twice a day, for 19 23 days. At the baseline study visit, they will get a supply of the study drug tablets and instructions for taking them. Participants will keep a medicine diary to serve as a memory aid for taking medicine and reporting any side effects that they may experience.

Participants will have 8 or 9 study visits over about 40 days. The number of visits depends on which group the person is assigned to. All visits will take place at the NIH Clinical Center. Participants will fast before study visits.

The baseline visit will last about 2 3 hours. There will be 3-4 long visits that will last for about 12 hours. The other 4-5 visits will last about 1 hour.

During all study visits, screening procedures will be repeated. During long visits, an intravenous (IV) line will be inserted into an arm vein with a needle. It will be used to take blood.

DETAILED DESCRIPTION:
Rifapentine (RPT) is a long-acting rifamycin that can be used weekly with isoniazid (INH) as a first-line regimen in the treatment of latent tuberculosis infection (LTBI). Although this regimen offers several potential benefits, the use of weekly RPT plus INH is not currently recommended in adults infected with human immunodeficiency virus (HIV) on antiretroviral therapy (ART) due to limited evidence on drug interactions with antiretrovirals (ARVs).1Darunavir boosted with cobicistat (DRV/c) comprises part of alternative treatment regimens recommended for the treatment of HIV.2However, drug interactions between these ARV agents and RPT are of concern. Thus, the purpose of this study is to determine the effects of concomitant RPT and INH administration on the steady state PK of DRV/c.

This is an open-label, fixed sequence, intrasubject drug-drug interaction study designed to evaluate the steady state PK of DRV/c with coadministration of once weekly RPT and INH given at doses used to treat LTBI. Arm B will be comprised of two phases: (1) DRV/c once daily alone (days 1-4) and (2) DRV/c once daily + (RPT and INH) once weekly (days 5-19). Participants in Arm B will undergo periodic serial ARV PK blood draws on days 4, 14, and 19.

DRV/c PK parameters will be determined using non-compartmental methods. Cobicistat levels will only be assessed if DRV concentrations are significantly decreased. The following PK parameters will be compared between phases: area under the curve over the dosing interval, maximum plasma concentration, time to maximum plasma concentration, terminal half-life, apparent oral clearance, and minimum plasma concentration. Adverse events will be graded and recorded.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be considered eligible for this study only if all of the following criteria are met:

1. Ages 18 - 65 years
2. Weight greater than or equal to 45 kg and less than or equal to 120; BMI greater than or equal to 18.0 and <30
3. Judged to be healthy based on medical history, physical examination, vital signs, and clinical laboratory tests (liver function tests (AST, ALT, Tbili) greater than or equal to upper limit of normal [ULN], serum creatinine (SCr) less than or equal to ULN, CK less than or equal to 2X ULN, platelets (PLT) >150,0000/mm3, hemoglobin (Hgb) >11 g/dL), C-reactive protein (CRP) less than or equal to ULN)
4. Negative QuantiFERON-TB Gold test at screening
5. HIV-negative, as determined by standard serologic assays for HIV infection.
6. No laboratory evidence of active Hepatitis A, B, or C infection
7. Willing to abstain from alcohol consumption throughout the study period
8. Subject agrees to genetic testing and storage of specimens for future research
9. Negative serum or urine pregnancy test for females of child-bearing potential
10. For female subjects able to become pregnant (i.e., have not undergone surgical sterilization or are not postmenopausal), willingness to prevent pregnancy during the study period by:

    1. Practicing absolute abstinence from sexual contact or
    2. Committing to use of effective non-hormonal and/or barrier methods of birth control during any and all sexual encounters. Acceptable methods are as follows:

       * Condom, diaphragm, or cervical cap with a spermicide
       * Intrauterine device (IUD) without hormones
       * Male partner with a vasectomy

EXCLUSION CRITERIA:

A subject will be ineligible for this study if 1, or more, of the following criteria are met:

1. Known hypersensitivity to dolutegravir, darunavir, cobicistat, rifapentine and other rifamycin analogues, or isoniazid
2. History of type 1 hypersensitivity reaction to sulfonamides
3. History or presence of any of the following:

   1. Latent or active TB infection
   2. Gastrointestinal disease that is uncontrolled, requires daily treatment with medication, or would interfere with a subject s ability to absorb drugs (diarrhea, pancreatitis, peptic ulcer disease, etc.),
   3. Renal impairment (chronic renal insufficiency of any CKD stage, or acute renal failure not induced by drug therapy defined as GFR < 90 ml/min)
   4. Respiratory disease that is uncontrolled or requires daily treatment with medication (asthma, chronic obstructive pulmonary disease, etc.)
   5. Cardiovascular disease (hypertension [systolic blood pressure >140 mmHg or diastolic blood pressure > 90 mmHg], heart failure, arrhythmia, etc.)
   6. Metabolic disorders (diabetes mellitus, etc.)
   7. Hematologic or bleeding disorders (anemia, hemophilia, serious/major bleeding events, menorrhagia (female subjects), etc.)
   8. Immunologic disorders
   9. Hormonal or endocrine disorders
   10. Psychiatric illness that would interfere with his or her ability to comply with study procedures or that requires daily treatment with medication
   11. Seizure disorder, with the exception of childhood febrile seizures
   12. Malignancy, or
   13. Any other condition that may interfere with the interpretation of the study results, or not be in the best interest of the subject in the opinion of the investigator
4. Fasting total cholesterol >240 mg/dL or fasting triglycerides >240 mg/dL on 2 consecutive visits
5. Fasting glucose >125 mg/dL on 2 consecutive visits
6. Current participation in an onging investigational drug protocol or use of any investigational drug within 30 days (based on last dose received) prior to receipt of any study drugs/medications.
7. Therapy with any prescription, over-the-counter, herbal, or holistic medications, including hormonal contraceptives by any route, within 5 half-lives of the agent prior to receipt of any study medications will not be permitted with the following exception: Intermittent or short-course therapy (< 14 days) with prescription or over-the-counter medications, herbals, or holistic medications within the screening period prior to starting study drug may be permitted, and will be reviewed by investigators on a case-by-case basis for potential drug interactions. Receipt of influenza vaccination will be allowed prior to, during, and/or after the study
8. Inability to obtain venous access for sample collection
9. Inability to swallow whole capsules and/or tablets
10. Current breastfeeding
11. Drug or alcohol use that may impair safety or adherence
12. Use of nicotine-containing products, including cigarettes and chewing tobacco, nicotine patches, gum, electronic cigarettes, etc.
13. Organ or stem cell transplant recipient
14. Uncorrected and persistent electrolyte abnormalities (e.g., potassium, magnesium, and calcium)
15. Current alcohol abuse or alcohol dependence disorders (DSM-5 criteria)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Area-under-the-curve during the dosing interval of 0 to t (AUC0-t), maximum total plasma concentration (Cmax), time to maximum plasma concentration (t-max), terminal halflife (t1/2), apparent oral clearance (CL/F) | Days 4 14, and 19
  To assess the effects of once weekly administration of RPT and INH given at doses used for treating LTBI on the steady state PK of DRV/c

SECONDARY OUTCOMES:
AEs and abnormal laboratory values graded according to the Division of AIDS AE Table, laboratory measures: hepatic & renal function, lipids, complete blood count, creatine kinase & lipase | Day 34
  To assess the safety of coadministration of DRV/c with once weekly RPT and INH through documentation of adverse events (AE) according to the Division of AIDS AE table

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.Individual participant data will not reported or shared. The study team are the only individuals who have access to individual participant data. All data will be analyzed and reported in aggregate.

REFERENCES:
- [Background] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833
- [Derived] Brooks KM, George JM, Pau AK, Rupert A, Mehaffy C, De P, Dobos KM, Kellogg A, McLaughlin M, McManus M, Alfaro RM, Hadigan C, Kovacs JA, Kumar P. Cytokine-Mediated Systemic Adverse Drug Reactions in a Drug-Drug Interaction Study of Dolutegravir With Once-Weekly Isoniazid and Rifapentine. Clin Infect Dis. 2018 Jul 2;67(2):193-201. doi: 10.1093/cid/ciy082. PMID 29415190
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0112.html

DOCUMENTS (1):
  • Informed Consent Form (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT02771249/ICF_000.pdf